CLINICAL TRIAL: NCT02842424
Title: Ramipril Treatment of Claudication: Oxidative Damage and Muscle Fibrosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0139-16-ET; 00991 (Other: VAMC-IRB)
Record Dates: First submitted 2016-06-17; First posted 2016-07-22 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Ramipril; Angiotensin-converting enzyme; Claudication; Myopathy; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Muscular Diseases | interventions — Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ramipril Treatment (Experimental): 6 months treatment with the medication Ramipril
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — Ramipril therapy will start at 2.5mg/day for 1 week. Then 5mg/day for 1 week and will be increased to 10mg/day by the third week. The patients will stay on Ramipril 10mg/day for 22 weeks.
  Other Names: Altace

SUMMARY:
Peripheral artery disease (PAD) is a manifestation of atherosclerosis that produces progressive narrowing and occlusion of the arteries supplying the lower extremities. The most common clinical manifestation of PAD is claudication, i.e., a severe functional limitation identified as gait dysfunction and walking-induced leg muscle pain relieved by rest. The standard therapies for claudication include the medications cilostazol and pentoxifylline, supervised exercise therapy and operative revascularization. Recent data demonstrated that 24 weeks of treatment with the angiotensin-converting enzyme (ACE) inhibitor Ramipril produces improvements in the walking performance of patients with claudication that are higher than those of cilostazol and pentoxifylline and similar to those produced by supervised exercise therapy and operative revascularization. The mechanisms by which Ramipril therapy produces this impressive improvement in the functional capacity of claudicating patients remain unknown. The Investigators hypothesize that treatment of claudicating PAD patients with Ramipril will improve walking performance and quality of life by improving the myopathy of the gastrocnemius. Improved myopathy is a consequence of reduced oxidative damage, reduced TGF-β1 production by vascular smooth muscle cells and reduced collagen deposition in the affected gastrocnemius.

DETAILED DESCRIPTION:
This is an interventional study of PAD patients that exhibit claudication. The purpose of this study is to determine the potential mechanisms by which Ramipril vastly improves the walking performance of these patients. The study will be achieved through these specific aims:

Specific Aim #1: Test the hypothesis that Ramipril-mediated improvements of walking parameters among patients with PAD correlate with improvements in both the morphometrics and biochemistry of myofibers in the gastrocnemius of the impaired limb.

Specific Aim #2: Test the hypothesis that Ramipril-mediated improvements of walking parameters in patients with PAD correlate with reduced fibrotic events in small vessels and microvasculature, in association with reduced generalized collagen deposition and improved tissue oxygenation, in the gastrocnemius of the impaired limb.

Specific Aim #3: Using adult human arterial smooth muscle cells (AHASMC), in vitro, the Investigators will test the hypothesis that the ACE inhibitor Ramipril, which acts as an antagonist of Angiotensin II type 1 receptor (ART1) stimulation by reducing tissue Angiotensin II (Ang II), impedes a mechanism in which Ang II stimulation of ART1 and exposure to hypoxia enhance proliferation of AHASMC and their production of TGF-β1 and collagen, via stimulation of phosphoinositide-3-kinase signaling and suppression of phosphatase and tensin homologue, a master regulator of cell growth.

If the above hypotheses are correct, Aims #1 and #2 will demonstrate for the first time that therapy with Ramipril improves the walking performance and quality of life of claudicating PAD patients by improving the myopathy in skeletal muscle of the ischemic lower limbs. The work in Aim #3 will determine the pathways by which hypoxia and Angiotensin II cooperate to induce myopathy in the ischemic muscle. Specific agents targeting these pathways could become new treatments for claudication and for the more advanced stages of PAD characterized by leg rest pain and gangrene.

ELIGIBILITY:
Inclusion Criteria:

1. A positive history of chronic claudication,
2. Exercise-limiting claudication established by history and direct observation during a screening walking test administered by the evaluating vascular surgeon,
3. Arterial occlusive disease per ankle Brachial index measurements and/or other imaging modalities,
4. Stable blood pressure regimen, stable lipid regimen, stable diabetes regimen and risk factor control for 6 weeks.

Exclusion Criteria:

1. Rest pain or tissue loss due to PAD (Fontaine stage III and IV),
2. acute lower extremity ischemic event secondary to thromboembolic disease or acute trauma,
3. Walking capacity significantly limited by conditions other than claudication including leg (joint/musculoskeletal, neurologic) and systemic (heart, lung disease) pathology,
4. Current use of either ACE inhibitors or angiotensin II receptor blockers,
5. Chronic kidney disease with estimated Glomerular Filtration Rate < 30 ml/min/1.73 m2,
6. History of bilateral severe renal artery stenosis and 7) History of angioedema related to previous ACE-inhibitor treatment or known hypersensitivity to ramipril or other ACE inhibitors.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-02-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Absolute Claudication Distance | 6 months
  Maximum walking distance in meters per Gardner protocol

SECONDARY OUTCOMES:
6-minute Walking Distance | 6 months
  Maximum Distance in meters the patient can walk in 6 minutes on a flat, hard surface
Initial Claudication Distance | 6 months
  The distance in meters the patient can walk before he experiences claudication pain, per Gardner protocol
Average Daily Steps Taken | 6 months
  Monitored with an accelerometer at home
Quality of life measured by the Walking Impairment Questionnaire | 6 months
  There are 14 questions across three categories of walking distance, walking speed and stair climbing. The WIQ is graded on a scale of 0-4; 0 represents no difficulty; 4 represents inability to walk. 0 score represents no difficulty, 1 score is slight difficulty, 2 score is some difficulty, 3 score is much difficulty, 4 score is unable to complete the task in question.
Quality of life measured by the Medical Outcomes Study Short Form 36 Healthy Survey | 6 months
  - (The Short Form 36 Health Survey Questionnaire) has 8 scale (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health) that measures quality of life. The SF-36 scoring ranges from 0-100. Higher scores indicate better health; lower scores indicate more disability
Leg biomechanics measured as Vertical ground reaction force | 6 months
  measured as Vertical ground reaction force
Leg hemodynamics measured as Ankle Brachial Index (ABI) | 6 months
  Ratio of the blood pressure at the level of the ankle to the blood pressure at the level of the arm
Leg hemodynamics | 6 months
  measured as Calf blood flow via contrast-enhanced ultrasound
Leg hemodynamics measured as Calf blood flow via stress ABI testing | 6 months
  measured as Calf blood flow via stress ABI testing
Leg hemodynamics measured as Calf muscle hemoglobin oxygen saturation | 6 months
  Measured with Near Infrared Spectroscopy
Myofiber Mitochondrial Respiration, measured by polarography | 6 months
  measured by polarography
Muscle Mitochondrial Function, measured by spectrophotometry | 6 months
  measured by spectrophotometry
Myofiber Oxidative Damage | 6 months
  Myofiber content of HNE adducts and protein carbonyls
Myofiber Morphology, Cross-Sectional Area | 6 months
  Area in square microns, measured by immunofluorescence microscopy
Myofiber Morphology, Roundness | 6 months
  Measured as ratio of major axis in microns to minor axis in microns
Myofiber Morphology, Solidity | 6 months
  Measured as the ratio of myofiber area in square microns to the area of a fitted convex hull in square microns
Muscle Fibrosis, Muscle TGF-β1 | 6 months
  Measured as the sum of the products of mean pixel intensity (in gray scale units) and area (in square microns) of each TGF-β1 labeled event divided by the total area (in square microns) of the tissue sample analyzed. Measured by immunofluorescence microscopy.
Muscle Fibrosis, Total collagen deposited. | 6 months
  Measured as the area-weighted mean pixel intensity (in gray scale units) of all the collagen labeled events per tissue sample. Measured by bright-field microscopy.
Microvascular Fibrosis, Capillary wall thickness. | 6 months
  Measured in microns by immunofluorescence microscopy of vessels labeled for collagen.
Capillary density. | 6 months
  Number of capillaries per unit area (in square microns) of the tissue sample analyzed.
Serum biomarker of fibrosis, serum procollagen type I c-peptide in picograms of peptide per ml | 6 months
  serum procollagen type I c-peptide in picograms of peptide
Serum biomarker of fibrosis, serum procollagen type III n-terminal peptide in picograms of peptide per ml | 6 months
  serum procollagen type III n-terminal peptide in picograms of peptide per ml
Plasma biomarker of fibrosis, plasma TGF-β1 in picograms per ml | 6 months
  plasma TGF-β1 in picograms per ml

CONTACTS AND LOCATIONS:
Overall Officials: Iraklis I Pipinos, MD, Principal Investigator — University of Nebraska; George P Casale, PhD, Principal Investigator — University of Nebraska
Locations (1):
- VA Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No